CLINICAL TRIAL: NCT04083417
Title: A Randomized Controlled Clinical Trial of Streptococcus Group A-negative Acute Tonsillitis in Primary Health Care - a Comparison of Phenoxymethylpenicillin and No Antibiotic Treatment
Brief Title: Sore Throat in Primary Care - a Comparison of Phenoxymethylpenicillin and No Antibiotic Treatment
Acronym: SANT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Katarina Hedin (Other Government)
Collaborators: Umeå University (Other); Linkoeping University (Other Government); Lund University (Other); Region JÃ¶nkÃ¶ping County (Unknown)
Responsible Party: Sponsor-Investigator, Katarina Hedin, Adjunct professor, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-000756-34
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Sore Throat; Tonsillitis
Keywords: sore throat; tonsillitis; randomized controlled trial; primary care; phenoxymethylpenicillin
MeSH Terms: conditions — Pharyngitis; Tonsillitis | interventions — Penicillin V

STUDY DESIGN:
Intervention Model Description: Randmization to antibiotic treatment or no antibiotic treatment
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenoxymethylpenicillin group (Active Comparator): Patients randomized to oral phenoxymethylpenicillin 1000 mg three times daily for ten days
  Interventions: Drug: Phenoxymethylpenicillin
- No antibiotic treatment group (Experimental): Patients randomized to no antibiotic treatment
  Interventions: Other: No antibiotic treatment

INTERVENTIONS:
Drug: Phenoxymethylpenicillin — tablet PcV 1000 mg x 3 for 10 days
  Other Names: Penicillin V (PcV)
  Arms: Phenoxymethylpenicillin group
Other: No antibiotic treatment — No prescription of antibiotics
  Arms: No antibiotic treatment group

SUMMARY:
Sore throat is the second most common cause of antibiotic prescribing in primary care in Sweden. Guidelines for sore throat focus on identifying people with sore throat where there are 3 and 4 specified criteria and where near patient tests identify group A streptococci (GAS). In these cases, phenoxymethylpenicillin is recommended.

Studies that have identified microorganisms in sore throat show that there are other bacteria and viruses than GAS, that give similar symptoms and that sometimes no microorganism is trapped despite pronounced symptoms. In recent years, a bacterium F. necrophorum has been identified, which is found in increased incidence of sore throat, but it is also found in healthy individuals. In clinical practice, many patients are treated with penicillin even if GAS is not captured. This may be because the doctor perceives the patient as sick or because other bacteria are not caught with a near patient test which causes the doctor to treat anyway.

The specific aims are to in patients with GAS-negative sore throat and 3 and 4 criteria, aged 15 years and older in primary care, study whether phenoxymethylpenicillin treatment shortens the duration of the disease, reduces the symptom intensity and sickness absence, and investigates the importance of other microorganisms than GAS in sore throat.

The study is a randomized controlled trial in which patients with sore throat are randomized to phenoxymethylpenicillin 3 times daily for 10 days or to no antibiotic therapy. There will also be and a reference group with severe (Centor score 3-4), GAS-positive acute tonsillitis.

Blood samples for inflammatory and immunological response to infections are taken. Throat samples for culture of F. necrophorum and streptococcal groups C and G, as well as polymerase chain reaction (PCR) analysis for bacteria and viruses are also taken at inclusion and at follow-up.

The outcome will be followed in a patient diary for 10 days and at a return visit after 18-24 days where the clinical outcome is asked for and where the blood- and throat samples are repeated.

Follow-up will also takes place via e-mail after 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

' Centor score 3-4: absence of cough, anamnestic fever (temperature >38.5°C), tender cervical lymphadenitis, and tonsillar exudates (one or both tonsils)

* Duration of symptoms < 8 days
* Rapid antigen detection test for GAS taken and negative
* Willing and able to give informed consent. Subjects under 18 years of age must in addition have the consent from both parents/caretakers

Exclusion Criteria:

* Ongoing antibiotic treatment
* Known or suspected allergies to phenoxymethylpenicillin
* Suspicion of peritonsillar abscess or indication for admittance.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Differences in number of days from inclusion to resolution of symptoms | 10 days after inclusion
  Differences between the randomized groups. Symptom resolution is defined as the first day the item sore throat and difficulty swallowing is scored less than moderately bad

SECONDARY OUTCOMES:
Proportions of patients with symptom resolution at each of the days 2 through 10. | up to 10 days after inclusion
The number of days from inclusion to symptom resolution of the individual items of sore throat symptoms. | 10 days after inclusion
Differences in number of days from inclusion to the day the patient can put up with the pain. | up to 10 days after inclusion
The possible change in the self-reported items of symptoms on the rating scale for each of the days 2 through 10 and describe the break through day for improvement | up to between 10 days after inclusion
  The rating is on a 7-point Likert scale 0=no symptoms, 1= very little, 2=slight, 3=moderately bad, 4=bad, 5=very bad, 6=as bad as it could be.
The number of days the patient needs to stay at home from work/school | 10 days after inclusion
Proportion of patients with future episodes of sore throat | 30 days and 3 months after inclusion
Proportion of patients at follow up with eradication of each of the potential pathogens found. | between 18 up to 24 days
  Bacteriological eradication
The number of adverse events | 3 months after inclusion
Description of patient characteristics and outcomes in the drop-out group. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Hedin, Ass Prof, Principal Investigator — Region Jönköping County
Locations (6):
- Sweden (6):
  - Vårdcentralen Rosenhälsan, Jönköping
  - Vårdcentralen Kärna, Linköping
  - Vårdcentralen Lundbergsgatan, Malmo
  - Mariehems hälsocentral, Umeå
  - Ålidhems hälsocentral, Umeå
  - Vårdcentralen Skärvet, Vaxjo

IPD SHARING:
Plan to Share IPD: No